CLINICAL TRIAL: NCT05524714
Title: Plasmakinetics of Micellar Solubilized Xanthohumol in Metabolically Healthy Men and Women
Brief Title: Plasma Appearance of Xanthohumol in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bonn (Other)
Collaborators: University of Hohenheim (Other)
Responsible Party: Principal Investigator, Prof. Dr. Sarah Egert, Prof. PhD, University of Bonn
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: XN BV
Record Dates: First submitted 2022-08-15; First posted 2022-09-01 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Plasmakinetics of Xanthohumol
Keywords: Polyphenols; Hops; Bioavailability; Xanthohumol; Plasma Kinetics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- solubilized Xanthohumol low dose (Experimental): single dose of 86 mg micellar solubilized Xanthohumol
  Interventions: Dietary Supplement: solubilized Xanthohumol low dose
- solubilized Xanthohumol high dose (Experimental): single dose of 172 mg micellar solubilized Xanthohumol
  Interventions: Dietary Supplement: solubilized Xanthohumol high dose
- native Xanthohumol low dose (Active Comparator): single dose of 86 mg native Xanthohumol
  Interventions: Dietary Supplement: native Xanthohumol low dose
- native Xanthohumol high dose (Active Comparator): single dose of 172 mg native Xanthohumol
  Interventions: Dietary Supplement: native Xanthohumol high dose

INTERVENTIONS:
Dietary Supplement: solubilized Xanthohumol low dose — single administration of 2 soft gelatine capsules each containing 43 mg micellar solubilized Xanthohumol and 2 soft gelatine capsules containing only micelles
  Arms: solubilized Xanthohumol low dose
Dietary Supplement: solubilized Xanthohumol high dose — single administration of 4 soft gelatine capsules each containing 43 mg micellar solubilized Xanthohumol
  Arms: solubilized Xanthohumol high dose
Dietary Supplement: native Xanthohumol low dose — single administration of 2 hard gelatine capsules each containing 43 mg native Xanthohumol and 2 hard gelatine capsules containing silicon dioxide
  Arms: native Xanthohumol low dose
Dietary Supplement: native Xanthohumol high dose — single administration of 4 hard gelatine capsules each containing 43 mg native Xanthohumol
  Arms: native Xanthohumol high dose

SUMMARY:
The aim of this study is to investigate the rate and extend of the plasma appearance of native Xanthohumol and Xanthohumol integrated into micelles in healthy men and women. Therefore, participants consume capsules with either 86 or 172 mg of native Xanthohumol or Xanthohumol integrated into micelles. In an observation period of 24 hours, Xanthohumol and its major metabolites are analyzed in plasma.

DETAILED DESCRIPTION:
In a crossover design, 6 healthy young men and 6 healthy young women participate in 4 Xanthohumol interventions with either 86 or 172 mg native or micellar solubilized Xanthohumol. During an observation period of 24 hours, Xanthohumol and its major metabolites Isoxanthohumol, 8- and 6-Prenylnaringenin are analyzed in plasma. Each intervention will be separated by a wash-out period of 14 days. Typical plasmakinetic analyses (Cmax, tmax, AUC, t1/2, bioavailability) will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 18,5 - 24,9 kg/m2
* metabolically healthy
* written consent

Exclusion Criteria:

* smoking
* low or high blood pressure
* dyslipidemia
* insulin resistance or diabetes mellitus type 1 or type 2
* gastrointestinal diseases (e.g. food intolerances or allergies)
* liver, kidney and/or thyroid diseases
* hepatitis B or C, HIV Infection
* chronic inflammatory diseases
* disordered eating
* psychological diseases
* alcohol and/or drug abuse
* veganism or unbalanced diets
* use of medication
* pregnancy or lactating
* participation in another intervention study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Systemic exposure to Xanthohumol | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9 and 24 hours post dose
  Mean area under the curve (AUC) of plasma concentration vs. time of total Xanthohumol (nmol/L*h)
Cmax Xanthohumol | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9 and 24 hours post dose
  Mean maximum plasma concentration of total Xanthohumol (nmol/L)
tmax Xanthohumol | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9 and 24 hours post dose
  Time to reach maximum plasma concentration of total Xanthohumol [h]
Oral bioavailability Xanthohumol | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9 and 24 hours post dose
  Minimum bioavailable amount of the ingested compound (%)

SECONDARY OUTCOMES:
Systemic exposure to Xanthohumol glucuronides | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9 and 24 hours post dose
  Mean area under the curve (AUC) of plasma concentration vs. time of Xanthohumol glucuronides (nmol/L*h)
Systemic exposure to Xanthohumol sulfates | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9 and 24 hours post dose
  Mean area under the curve (AUC) of plasma concentration vs. time of Xanthohumol sulfates (nmol/L*h)
Systemic exposure to free Xanthohumol | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9 and 24 hours post dose
  Mean area under the curve (AUC) of plasma concentration vs. time of free Xanthohumol (nmol/L*h)
Cmax Xanthohumol glucuronides | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9 and 24 hours post dose
  Mean maximum plasma concentration of Xanthohumol glucuronides (nmol/L)
Cmax Xanthohumol sulfates | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9 and 24 hours post dose
  Mean maximum plasma concentration of Xanthohumol sulfates (nmol/L)
Cmax free Xanthohumol | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9 and 24 hours post dose
  Mean maximum plasma concentration of free Xanthohumol (nmol/L)
tmax Xanthohumol glucuronides | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9 and 24 hours post dose
  Time to reach maximum plasma concentration of Xanthohumol glucuronides [h]
tmax Xanthohumol sulfates | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9 and 24 hours post dose
  Time to reach maximum plasma concentration of Xanthohumol sulfates [h]
tmax free Xanthohumol | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9 and 24 hours post dose
  Time to reach maximum plasma concentration of free Xanthohumol [h]

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Egert, Prof PhD, Principal Investigator — University of Bonn
Locations (1):
- University of Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No